CLINICAL TRIAL: NCT03766061
Title: Onlay Mesh Hernioplasty Vs Sublay Mesh Hernioplasty for Paraumbilical Hernia Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Services Hospital, Lahore (Other Government)
Responsible Party: Principal Investigator, Dr. SamiUllah, Principle investigator, Services Hospital, Lahore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: s8
Record Dates: First submitted 2018-07-13; First posted 2018-12-05 (Actual); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Paraumbilical Hernia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Onlay Mesh Hernioplasty (Active Comparator): In this group patients with paraumbilical hernia are treated with onlay mesh hernioplasty in which we placed mesh on the anterior rectus sheath
  Interventions: Procedure: Onlay mesh Hernioplasty
- Sublay Mesh Hernioplasty (Active Comparator): In this group patients with paraumbilical hernia are treated with sublay mesh hernioplasty in which we placed mesh in the retromuscular space
  Interventions: Procedure: Sublay Mesh Hernioplasty

INTERVENTIONS:
Procedure: Onlay mesh Hernioplasty — Patients with paraumblical hernia are treated with onlay mesh hernioplasty in which mesh is placed on anterior rectus sheath
  Arms: Onlay Mesh Hernioplasty
Procedure: Sublay Mesh Hernioplasty — Patients with paraumblical hernia are treated with sublay mesh hernioplasty in which mesh is placed in retromuscular space
  Arms: Sublay Mesh Hernioplasty

SUMMARY:
It is a randomized controlled trial in which we are comparing onlay mesh hernioplasty with sublay mesh hernioplasty for paraumbilical hernia.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes and age 20 years and above with paraumblical hernia Defect size 3 to 6cm in greatest diameter

Exclusion Criteria:

* defect size less than 3cm or greater than 6 cm in greatest diameter Obstructed or strangulated hernia Uncontrolled diabetes

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
Percentage of patients presenting with recurrence of hernia | 8 months
  Recurrence (defined as appearance of swelling in operative site with positive cough impulse) of hernia after surgery

SECONDARY OUTCOMES:
Postoperative pain from score 1 to 10 | 3 days
  Postoperative pain measured with visual analog score after surgery with 1 being the minimum and 10 being the maximum
Hospital Stay duration in days | 1 week
  hospital stay (duration of patient from surgery to discharge) after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Mahmmood Ayyaz, mbbs, fcps, Study Director — Services Hospital, Lahore
Locations (1):
- Services hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided